CLINICAL TRIAL: NCT03347656
Title: Effects of Mobility Dose on Discharge Disposition in Critically Ill Stroke Patients
Status: Completed | Type: Observational
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Massachusetts General Hospital (Other); Technical University of Munich (Other)
Responsible Party: Principal Investigator, Balachundhar Subramaniam, Professor of Anesthesia, Beth Israel Deaconess Medical Center
Other Study IDs: 2017P000528
Record Dates: First submitted 2017-11-13; First posted 2017-11-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Sarcopenia; Stroke, Acute; Muscle Weakness; Critical Illness
Keywords: Mobilization Therapy; Clitical Illness; Stroke; Intensive Care; Functional Mobility; Quality of Life
MeSH Terms: conditions — Sarcopenia; Stroke; Muscle Weakness; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary aim of the study is to assess the mobility dose in neurocritical care patients with ischemic stroke or intracranial hemorrhage and its effects on discharge disposition and patient outcomes. The investigators hypothesize that patients' mobilization dose in the intensive care unit (ICU) predicts discharge disposition, 90 day Barthel Index and other outcomes like muscle wasting (expressed as decrease in rectus femoris cross sectional area (RF-CSA) in the paretic and non-paretic limb measured by bedside ultrasound), and ICU length of stay (LOS).

DETAILED DESCRIPTION:
The investigators have previously developed and validated the Surgical Intensive Care Unit Optimal Mobilization Score (SOMS), an algorithm to guide and facilitate early mobilization to advance mobility of surgical intensive care unit patients (NCT01363102). In addition, the investigators have established the use of bedside ultrasound technology to quantify cross sectional area of the rectus femoris muscle, which allows an objective, user-independent quantification of muscle wasting (NCT02270502).

This is a prospective, observational study to observe the relation between mobility dose, muscle wasting and patient outcomes in critically ill stroke patients.

Patients will be enrolled within 48 hours of ICU admission. The investigators will measure the dose of activity, that is duration and intensity of mobilization in critically ill patients with ischemic stroke and intracerebral hemorrhage. By mobility "dose" the investigators are referring to all provider-directed activities (by nursing, and physical therapists) meant to enhance the patient's mobility level. The investigators take into account mobility "dose", defined as a function of both the mobility level (e.g., sitting at the edge of the bed, ambulating) as well as its duration. Of note, there is so far no published data available that describes patients' mobility "dose" in such an integrative, semi-quantitative fashion.

The investigators use the existing mobility intensity quantification tool (MQS) (NCT03196960) and test the hypotheses that mobilization dose predicts muscle wasting in critically ill stroke patients, adverse hospital discharge disposition as well as 90 day Barthel Index. The investigators will apply hierarchical testing to evaluate the association between mobilization dose and discharge disposition as well as 90-day Barthel Index.

The Mobilization Quantification Score (MQS) is a composition of the validated ICU mobility score (SOMS), a 0 to 10 value scale that measures the mobility milestones in critically ill patients, multiplied by a for each level previously defined time unit (5 or 30 minutes correspond to one unit depending on mobilization level).

In order to capture the muscle status at ICU admission, determined by the first bedside ultrasound of the rectus femoris muscle after enrollment, and the change in rectus femoris muscle diameter throughout stay, the investigators will conduct repetitive measurements of the cross sectional area of the rectus femoris muscles (RF-CSA) of both legs. This longitudinal setting will allow to investigate muscle wasting due to immobilization and other severe illness related factors in the paretic and non-paretic limb.

The investigators will conduct a scheduled phone call 30 days and 90 days after hospital discharge by getting in contact with either the patient or a family member to obtain follow-up data. This conversation will include questions that allow to identify the Barthel Index at 30 days, the Barthel Index and GOS-E score at 90 days, and if the patient has been readmitted to a hospital within 30 days of hospital discharge and mortality.

Discharge disposition is defined as discharge to facilities providing long-term care assistance for daily activities, including nursing homes and skilled nursing facilities, hospice at the patient's home, hospice in a health care facility; or in-hospital mortality. The Barthel Index is a measure of functional disability originally designed to evaluate progress of rehabilitation in patients with stroke and neuromuscular disease. The GOS-E (Extended Glasgow Outcome Scale) is a global scale for functional outcome that rates patient status into eight categories: Dead Vegetative State, Upper and Lower Severe Disability, Upper and Lower Moderate Disability, Upper and Lower Good Recovery.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years and older
* Admitted to the neurological intensive care service within the past 48 hours
* an expected ICU length of stay of at least 48h
* New onset ischemic stroke or non-traumatic intracerebral hemorrhage
* Baseline functional independence: Barthel-Index of 70 or above 2 weeks before admission (obtained retrospectively from patient or proxy)

Exclusion Criteria:

* Transfers from other institutions (hospitals, long-term rehabilitation facilities, skilled nursing facilities) with a stay >48h at the outside institution
* absence of lower extremities
* not committed to full support
* exclusive or clinically predominant posterior circulation ischemic stroke
* subarachnoid hemorrhage, subdural and epidural hemorrhage

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: critically ill stroke patients recovering in the neurological intensive care unit
Sampling Method: Non-Probability Sample
Enrollment: 164 (Actual)
Dates: Start 2017-10-12 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Adverse Hospital Discharge Disposition | patient will be followed until hospital discharge; assessed at hospital discharge; expected between study day 3 and 30
  Adverse hospital discharge is defined as discharge to facilities providing long-term care assistance for daily activities, including nursing homes and skilled nursing facilities, hospice at the patient's home, hospice in a health care facility, or in-hospital mortality.
90 day Barthel Index (hierarchical testing) | 90 days post discharge from hospital (collected through follow up phone call)
  The Barthel Index is a measure of functional disability originally designed to evaluate progress of rehabilitation in patients with stroke and neuromuscular disease.

SECONDARY OUTCOMES:
Rectus Femoris Muscle Cross Sectional Area Rectus Femoris Muscle Cross Sectional Area | will be measured at least twice (on day of enrollement and before discharge); if stay longer than one week, ultrasound will be performed weekly (every 7 days); expected total time period of 3 to 30 days
  Rectus femoris cross sectional area will be measured by bedside ultrasound, raw numbers as well as change over time will be respected
30 day Barthel Index | 30 days post discharge from hospital (collected through follow up phone call)
  The Barthel Index is a measure of functional disability originally designed to evaluate progress of rehabilitation in patients with stroke and neuromuscular disease.
Neurological ICU length of stay | admission until discharge from neurological ICU; an expected 3 to 20 days
  number of days patient stays on the neurological ICU
Neurological ICU length of stay until discharge readiness | admission until discharge readiness from neurological ICU; an expected 3 to 20 days
  number of days patient stays on the neurological ICU until time point from which patient is stable for discharge from ICU
hospital length of stay | admission until discharge from hospital: patient will be followed until discharge from hospital; an expected 3 to 30 days
  number of days patients stays in hospital during index admission
FIM Score at ICU discharge | assessed at discharge from neurological ICU; expected between study day 3 and 20
  Functional independence measure score in the domains transfer and locomotion at ICU discharge
Days on sedation | during hospital stay; an expected 0 to 30 days
  number of days patient receives sedatives
mortality | during ICU stay, hospital stay or within the 30day or 90day follow up period (follow up data collected through phone call
  we will distinguish between ICU mortality, hospital mortality and mortality within 30 or 90 days after discharge from hospital
ICU readmission | during hospital stay; expected to be assessed between study day 3 and 30
  readmission to the ICU after discharge from ICU but within hospital stay
30-day hospital readmission | 30 days after discharge from hospital, obtained through follow up phone call
  readmission to a hospital within 30 days after discharge from index stay
90-day GOS-E (Extended Glasgow Outcomes Scale) | obtained 90 days after discharge from hospital through follow up phone call
  The GOS-E is a global scale for functional outcome that rates patient status into eight categories: Dead Vegetative State, Upper and Lower Severe Disability, Upper and Lower Moderate Disability, Upper and Lower Good Recovery
Total costs of care | during hospital stay
  total costs of care
Falls | during hospital stay; expected to be assessed between study day 3 and 30
  number of falls
Delirium-free days | CAM-ICU will be evaluated daily during hospital stay; an expected 0 to 30 days
  defined by CAM-ICU (Confusion Assessment Method)

CONTACTS AND LOCATIONS:
Overall Officials: Balachundhar Subramaniam, MD, MPH, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (3):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deconess Medical Center, Boston, Massachusetts
- Klinikum rechts der Isar of Technische Universität München, Munich, Bavaria, Germany

REFERENCES:
- [Background] Schaller SJ, Anstey M, Blobner M, Edrich T, Grabitz SD, Gradwohl-Matis I, Heim M, Houle T, Kurth T, Latronico N, Lee J, Meyer MJ, Peponis T, Talmor D, Velmahos GC, Waak K, Walz JM, Zafonte R, Eikermann M; International Early SOMS-guided Mobilization Research Initiative. Early, goal-directed mobilisation in the surgical intensive care unit: a randomised controlled trial. Lancet. 2016 Oct 1;388(10052):1377-1388. doi: 10.1016/S0140-6736(16)31637-3. PMID 27707496
- [Background] Mueller N, Murthy S, Tainter CR, Lee J, Riddell K, Fintelmann FJ, Grabitz SD, Timm FP, Levi B, Kurth T, Eikermann M. Can Sarcopenia Quantified by Ultrasound of the Rectus Femoris Muscle Predict Adverse Outcome of Surgical Intensive Care Unit Patients as well as Frailty? A Prospective, Observational Cohort Study. Ann Surg. 2016 Dec;264(6):1116-1124. doi: 10.1097/SLA.0000000000001546. PMID 26655919
- [Background] Lee JJ, Waak K, Grosse-Sundrup M, Xue F, Lee J, Chipman D, Ryan C, Bittner EA, Schmidt U, Eikermann M. Global muscle strength but not grip strength predicts mortality and length of stay in a general population in a surgical intensive care unit. Phys Ther. 2012 Dec;92(12):1546-55. doi: 10.2522/ptj.20110403. Epub 2012 Sep 13. PMID 22976446
- [Background] Kasotakis G, Schmidt U, Perry D, Grosse-Sundrup M, Benjamin J, Ryan C, Tully S, Hirschberg R, Waak K, Velmahos G, Bittner EA, Zafonte R, Cobb JP, Eikermann M. The surgical intensive care unit optimal mobility score predicts mortality and length of stay. Crit Care Med. 2012 Apr;40(4):1122-8. doi: 10.1097/CCM.0b013e3182376e6d. PMID 22067629
- [Background] Sainsbury A, Seebass G, Bansal A, Young JB. Reliability of the Barthel Index when used with older people. Age Ageing. 2005 May;34(3):228-32. doi: 10.1093/ageing/afi063. PMID 15863408
- [Background] Inouye SK, van Dyck CH, Alessi CA, Balkin S, Siegal AP, Horwitz RI. Clarifying confusion: the confusion assessment method. A new method for detection of delirium. Ann Intern Med. 1990 Dec 15;113(12):941-8. doi: 10.7326/0003-4819-113-12-941. PMID 2240918
- [Background] Wilson JT, Pettigrew LE, Teasdale GM. Structured interviews for the Glasgow Outcome Scale and the extended Glasgow Outcome Scale: guidelines for their use. J Neurotrauma. 1998 Aug;15(8):573-85. doi: 10.1089/neu.1998.15.573. PMID 9726257